CLINICAL TRIAL: NCT04581811
Title: Prolonged Prone Positioning for COVID-19-induced Acute Respiratory Distress Syndrome (ARDS): A Pilot Study
Brief Title: Prolonged Prone Positioning for COVID-19-induced Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Page, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300005979
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: ARDS; Covid19; Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged Proning Arm (Experimental): Patients will receive 24 hours in the prone position followed by 8 hours in the supine position for the duration of the study
  Interventions: Other: Prolonged Proned Positioning
- Traditional Proning Arm (Active Comparator): Patients will receive standard 16 hour prone positioning followed by 8 hours in the supine position for the duration of the study
  Interventions: Other: Traditional Proning Arm

INTERVENTIONS:
Other: Prolonged Proned Positioning — Patients will be placed in the prone position for 24 hours followed by 8 hours supine for consecutive periods for the duration of the study period
  Arms: Prolonged Proning Arm
Other: Traditional Proning Arm — Patients will be placed in the prone position for 16 hours followed by 8 hours supine for consecutive periods for the duration of the study period
  Arms: Traditional Proning Arm

SUMMARY:
Prone positioning is one of the few therapies known to improve mortality in ARDS. Traditionally, patients are proned for 16 hours per 24 hour period. Some retrospective data suggests improvement may persist beyond 16 hours. We aim to perform a pilot study comparing traditional prone positioning to prolonged prone positioning in patients with COVID-induced ARDS.

ELIGIBILITY:
Inclusion Criteria:

Positive COVID test Endotracheal Intubation P:F <150 within 1hours of inclusion on at least 60% FiO2, 10cmH20 PEEP Treating physician plans to implement prone positioning imminently Housed in the UAB MICU.

Exclusion Criteria:

Pre-existing treatment limitation (e.g. DNR order) Prisoner Pregnant Female Children (<18 years old) Respiratory Failure felt to be caused primarily by something other than COVID-19 Mechanical ventilation for >48 hours prior to initiation of prone positioning Contraindication to proning Physician discretion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Page DB, Vijaykumar K, Russell DW, Gandotra S, Chiles JW, Whitson MR, Dransfield MT. Prolonged Prone Positioning for COVID-19-induced Acute Respiratory Distress Syndrome: A Randomized Pilot Clinical Trial. Ann Am Thorac Soc. 2022 Apr;19(4):685-687. doi: 10.1513/AnnalsATS.202104-498RL. No abstract available. PMID 34491885

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (14) | 62 (12) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Duration in Prone Position
Description: Time spent in the prone position of hours eligible for prone positioning
Time Frame: 96 hours
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Prolonged Proning Arm: Patients will receive 24 hours in the prone position followed by up to 8 hours in the supine position for the duration of the study
- Traditional Proning Arm: Patients will receive standard 16 hour prone positioning followed by up to 8 hours in the supine position for the duration of the study
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
hours | 56.6 (20.6) | 45.7 (20.8)

2. Secondary Outcome: Change in P:F Ratio
Description: Change in PaO2 on ABG to FiO2 ratio from immediately prior to initiation of prone positioning to end of study period
Time Frame: End of supine session on day 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Ratio | 46.6 (39.9) | 44.3 (63.7)

3. Secondary Outcome: Change in Drive Pressure
Description: Change in drive pressure from immediately prior to initiation of prone positioning to end of the study period
Time Frame: End of supine session on day 4
Measure: Mean (Standard Deviation); unit: cm H20
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
cm H20 | 0.16 (3.26) | 0.88 (4.95)

4. Secondary Outcome: Unplanned Extubations
Description: Number of unplanned extubations
Time Frame: End of supine session on day 4
Measure: Number; unit: Unplanned Extubations
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Unplanned Extubations | 0 | 1

5. Secondary Outcome: Pressure Ulcers
Description: Number of patients with pressure ulcers
Time Frame: End of supine session on day 4
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Participants | 1 | 0

6. Secondary Outcome: Line Displacement
Description: Number of displaced central venous line or arterial line
Time Frame: End of supine session on day 4
Measure: Number; unit: Central Venous or Arterial LineDislodged
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Central Venous or Arterial LineDislodged | 0 | 1

7. Secondary Outcome: Vent Free Days
Description: Number of days free from mechanical ventilation
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
days | 6.27 (9.15) | 5.81 (9.28)

8. Secondary Outcome: Mortality
Description: Mortality at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Participants | 14 | 15

9. Secondary Outcome: Rescue Interventions
Description: Patients in which new initiation of inhaled pulmonary vasodilators, ECMO
Time Frame: 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Participants | 0 | 1

10. Secondary Outcome: Tracheostomy
Description: Number of patients who have placement of tracheostomy
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Participants | 6 | 3

11. Secondary Outcome: ICU Free Days
Description: Number of days not in ICU
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
days | 4.35 (7.14) | 4.15 (7.52)

12. Secondary Outcome: S:F Ratio
Description: Ratio of SpO2 to FiO2
Time Frame: 96 hours
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
Number analyzed (Participants) | 26 | 26
Ratio | 1.70 (0.48) | 1.69 (0.52)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Prolonged Proning Arm | Traditional Proning Arm
All-Cause Mortality (participants affected / at risk) | 14/26 | 15/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04581811/Prot_SAP_000.pdf